CLINICAL TRIAL: NCT06920784
Title: Prismatic Adaptation for Cognitive Rehabiliation in Traumatic Brain Injury Patients
Brief Title: Prismatic Adaptation in Cognitive Rehabilitation
Acronym: PACoR-TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1791/CEL
Record Dates: First submitted 2025-02-04; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; prismatic adaptation; cognitive rehabilitation; serious games
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prismatic adaptation group (Experimental): Patients receiving treatment with prismatic lenses and serious games lasting 10 days over a span of 2 weeks, for 40 minutes each session. This training will be administered using a class I medical device SaMD (Software as a Medical Device) associated to prisms.
  Interventions: Device: PRISMATIC ADAPTATION; Device: Serious games
- Control group (Sham Comparator): patients receiving the same serious games for 10 days over a span of 2 weeks, withouth prismatic adaptation session.
  Interventions: Device: Serious games

INTERVENTIONS:
Device: PRISMATIC ADAPTATION — The experimental treatment includes a session of prismatic adaptation, in which patients, wearing priasmatic lenses, performs pointing exercises using an 11'' tablet. The visual target is represented by a black squares randomly presented in one of three spatial positions of the tablet's screen (in the centre of the screen or at 21° to the right or to the left space). Taking into account the type of lesion resulting from traumatic brain injury, the prismatic deviation induced by the lenses will be changed alternately from right to left. Then patients will wear rightward prism lenses for 5 days and leftward prism lenses for other 5 days. The prismatic deviation will be randomized.
  Following these prismatic adaptation, lasting 10 minutes, cognitive training with serious games will be performed, for the remaining 30 minutes.
  Arms: Prismatic adaptation group
Device: Serious games — patients receiving the same serious games for 10 days over a span of 2 weeks, withouth prismatic adaptation session.

SUMMARY:
The study aims to evaluate the effects of prismatic adaptation and then of a novel rehabilitation protocol that combines PA and Serious Games on cognitive and behavioural deficits in patients with traumatic brain injury , compared to a rehabilitation training without prismatic adaptation.

Moreover, this study aims to assess the impact of this rehabilitation protocol on functional cognitive outcomes.

Hypothesis Hypothesis 1 (H1): It is postulated that the utilization of Prismatic Adaptation Treatment (PAT) has a positive impact on the enhancement of cognitive outcome among patients suffering from TBI

Hypothesis 2 (H2): It is hypothesized that there will be discernible alterations in resting-state Electroencephalography (EEG) patterns between the initial assessment point (T0) and the subsequent measurement during the course of treatment (T1) in individuals diagnosed with TBI

Assessment times of outcome measures will be conducted before the experimental treatment (T0) and after the 10 rehabilitation sessions (T1).

Patients will be randomized into two groups:

1. Experimental group: Patients receiving treatment with prismatic lenses and serious games lasting 10 days over a span of 2 weeks, for 40 minutes each session.
2. Control group: patients receiving the same serious games for 10 days over a span of 2 weeks, withouth prismatic adaptation session.

Both groups will receive also the standard cognitive rehabilitation for the detected deficits, using paper and pen materials.

Each rehabiliation session will last aproximately 1 hour for 5 days a week for 2 weeks.

DETAILED DESCRIPTION:
Background Neurological diseases, such as Traumatic Brain Injury (TBI), represent a significant public health concern, with profound consequences on cognitive functions and overall quality of life. Attention, memory, and executive functions and behaviour are the cognitive domains usually impacted by TBI. Attentional and executive deficits represent the most pronounced cognitive deficits that impact every activity of daily life. As the field of neurorehabilitation continues to evolve, exploring innovative interventions becomes imperative. This study explores the efficacy of a promising modality, such as Prism Adaptation Treatment (PAT) on the cognitive rehabilitation of individuals with neuropsychological deficits following traumatic brain injury Prismatic lenses have shown potential in addressing visual and perceptual deficits and the association with cognitive rehabilitation with Serious Games could offer a dynamic cognitive rehabilitation means. Understanding the effects of these interventions would allow an enhancement of cognitive functions, providing valuable insights for developing effective and targeted rehabilitation strategies for patients. This research aims to contribute to the growing body of knowledge in neurorehabilitation and paves the way for improved therapeutic approaches to manage cognitive deficits following TBI.

Prismatic Lenses

Prism adaptation (PA) is a form of procedural learning in which the motor system adapts to new visuospatial coordinates imposed by prismatic lenses that displace the visual field horizontally. By introducing prisms that deviate the visual fields during movements, patients show initial pointing errors in the direction of the prism deviation. PA involves the progressive adaptation of patients to this visual distortion, gradually compensating for the initial errors over pointing trials. Removing prismatic lenses ends in a deviation of spatial attention towards the contralateral side. Studies on brain lesions unfold the neural circuitry underlying PA as a parieto-cerebellar network, where the anterior intraparietal sulcus detects the visual-motor misalignment produced by prisms, and the parieto-occipital sulcus invokes changes to correct the internal movement models.

The aftereffect, which can be observed in the spatial deviation of the motor actions in the direction opposite to the visual displacement imposed by the prisms, is a reliable measure of the degree and strength of the adaptation.

Prismatic lenses are typically adopted as a rehabilitative treatment for patients with visuospatial deficits, mainly Spatial Neglect (SN).

This being a common aftermath of TBI, hindering motor and cognitive rehabilitation and prolonging the length of stay. The effectiveness of prismatic lenses on TBI patients has been proved through 5-to-10 prismatic adaptation treatment (PAT) sessions, leading to an improvement of SN caused by the PA aftereffect, showcasing clinically meaningful progress across different SN severities.

The majority of observations in healthy samples shows that PA affects not only low-level sensory-motor processes, but also high-level cognitive functions, acting both on space representation and on other features interacting with this ability, such as visuospatial attention, time perception, number processing. This proves the potential of PA to neuromodulate brain excitability in a network ipsilateral to the deviation, resulting in a major impact on the related cognitive functions, leading to behavioral improvement coherent with the hemisphere modulated by the prism adaptation.

PA has also been proven to be associated with improved phonemic fluency performance in healthy subjects when the prisms are deviated to the left, rather than to the right, leading to an increase in word production and length. The former being consistent with the fact that left brain regions are associated with the dorsal language network, and, therefore, with phonemic fluency, as the latter is with frontal motor areas. Thus, those findings add up to the idea of a network activation induced by PA, that can bring a general improvement of cognitive functions.

It is important to acknowledge that further research is needed to fully understand the extent of prismatic lenses' effect on cognitive functions other than visuospatial abilities, since, even though PA needs active engagement in pointing task with prismatic lenses, the cognitive aftereffect is not fully explained by the sensorimotor adaptation.

Serious Games

Rehabilitation programs show that intensive and repetitive goal-oriented tasks can improve cognitive functions; however, implementing such an approach in a traditional rehabilitative protocol reduces patients' motivation to complete the exercises, perceived as boring and uninteresting due to their repetitive nature. On the other hand, Serious Games (SG) overcome this challenge, captivating patients thanks to a dynamic environment, useful to maintain the attentional threshold and sustain emotional processes through active, modern, and motivational tasks. Proven to be valuable tools in promoting brain plasticity, they improve cognitive skills, such as memory, attention, and perception.

Different studies assessed the crucial role of Serious Games in cognitive rehabilitation. For instance, a single-case study of a TBI patient, using 3D driving simulator to explore alterations in spatial and verbal memory, revealed stable short-term memory and a significant improvement in visuo-spatial memory learning, and in the verbal performance.

Enforcing Serious Games rehabilitation protocols in people with traumatic brain injury might be groundbreaking because it is still unknown whether the benefits of this training can be shifted to clinical settings and if games can improve cognitive functions engaged in daily activities.

Prismatic Adaptation (PA) and Cognitive Rehabilitation with Serious Games

Recently, the procedure of prismatic adaptation is digitized and the pointing movements are performed towards visual targets presented in various spatial positions of a tablet. Previous studies had showed that PA increases the excitability of a fronto-parietal network ispilateral to the side of spatial deviation. The following cognitive training, presented through serious games, harnesses the modulation power induced by the prisms to enhance the neurorehabiliation effect of cognitive training.

Oliveri et al. had evaluated, in a sample of 30 post stroke patients, the efficacy of the associations of PA and serious games specific for sustained and divided attention, working memory, interference control, inhibition and planning on cognitive rehabilitation. The results showed an enhancement in digit span forward, spatial span backward, attentional matrices, and Stroop tests in experimental group. Additionally, a notable correlation was observed between improved spatial span backward and improvements in activities of daily living, along with a reduction in anxiety levels.

There are no studies in the literature that have evaluating the effects of prismatic adaptation together with cognitive rehabilitation in traumatic brain injury patients. This study seeks to fill this gap, with the aim of offering a new rehabilitation opportunity that is easy and rapid to apply.

AIMS The study aims to evaluate the effects of prismatic adaptation through a novel rehabilitation protocol that combines PA and Serious Games on cognitive deficits in patients with traumatic brain injury, compared to usual rehabilitation training without prismatic adaptation, but considering the employment of serious games.

Moreover, this study aims to assess the impact of this rehabilitation protocol on behavioural and functional cognitive outcomes.

Hypothesis Hypothesis 1 (H1): It is postulated that the utilization of Prismatic Adaptation Treatment (PAT) has a positive impact on the enhancement of cognitive outcome among patients suffering from TBI

Hypothesis 2 (H2): It is hypothesized that there will be discernible alterations in resting-state Electroencephalography (EEG) patterns between the initial assessment point (T0) and the subsequent measurement during the course of treatment (T1) in individuals diagnosed with TBI.

STUDY DESIGN Experimental study, no-profit. All patients consecutively adimitted to Neurorehabiliation Unit of ICS Maugeri (Bari, Telese Sciacca, Pavia Italy) with Traumatic brain injury (TBI) will be enrolled in the study for 1 year, starting from May 1st.

PARTICIPANTS Inclusion Criteria

* Age >18 years
* Traumatic brain injury (TBI)
* Rancho Level of Cognitive Functioning (LCF) for TBI patients > 4
* Admission within 90 days from the onset

Exclusion Criteria

* Unilateral Spatial Neglect
* Aphasia
* Severe vigilance deficits
* Severe verbal comprehension deficits
* Motor deficits of both hands
* Previous neurological stroke
* Previous neurological disease
* Previous psychiatric disease
* Use of alcohol or drugs
* Severe visual deficits
* Premorbid dementia METHODS

All enrolled patients will be randomized into two groups, by a researcher not involved in this research:

1. Experimental group: Patients receiving treatment with prismatic lenses and serious games lasting 10 days over a span of 2 weeks, for 40 minutes each session. This training will be administered using a class I medical device SaMD (Software as a Medical Device) associated to prisms.

   The experimental treatment includes a session of prismatic adaptation, in which patients, wearing priasmatic lenses, performs pointing exercises using an 11'' tablet. The visual target is represented by a black squares randomly presented in one of three spatial positions of the tablet's screen (in the centre of the screen or at 21° to the right or to the left space). Taking into account the type of lesion resulting from traumatic brain injury, the prismatic deviation induced by the lenses will be changed alternately from right to left. Then patients will wear rightward prism lenses for 5 days and leftward prism lenses for other 5 days. The prismatic deviation will be randomized.

   Following these prismatic adaptation, lasting 10 minutes, cognitive training with serious games will be performed, for the remaining 30 minutes.

   The Serious Games aim to train sustained and divided attention, working memory, interference control, inhibition, and planning. Each game contains an adaptive difficulty mechanism that increases or decreases the difficulty according to the patient's performance:
   * sustained attention and monitoring task
   * visual search task
   * planning and switching
   * go-no go
   * visual working memory
   * math speed and digit working memory
   * semantic associations
2. Control group: patients receiving the same serious games for 10 days over a span of 2 weeks, withouth prismatic adaptation session.

Both groups will receive also the standard cognitive rehabilitation for the detected deficits, using paper and pen materials.

Each rehabiliation session will last aproximately 1 hour for 5 days a week for 2 weeks.

Assessment times of outcome measures will be conducted before the experimental treatment (T0) and after the 10 rehabilitation sessions, for both groups.

After post treatment assessment, both groups will continue standard cognitive rehabilitation treatment lasting 1 hour for 5 days a week.

All patients will receive standard motor rehabilitation and occupational therapy.

Neuropsychological primary outcome measure All patients will be assessed and enrolled immediately after the hospitalization.

Sample size determination The effect size to be expected is uncertain, as no study so far has implemented a combined intervention of PA and serious games for these patients. One previous study had assessed the efficacy of the same digital approach on the cognitive deficits in poststroke patients, enrolling 30 patients. In this study, the authors considered as outcome measures both neuropsychological tests and functional measures, such as Barthel Index.

Considering as the neuropsychological primary outcome the MoCA score, the investigators aim to achieve 90% power in a repeated-measures analysis of variance (a = 0.05, power (1-b) = 0.9) with condition as between-subject factor, and time as within-subject factor. Power calculations (using a Sample Size Calculator) indicate that a valid sample size of n = 25 per group will result in 90% statistical power if the effect is d = 0.5, which is in the medium-to-large range, considering a drop-out rate of 10%. This results in a total sample size of n = 50.

The investigators will enrol 50 patients with cognitive deficits following TBI. Each rehabilitation center is expected to enrol approximately 12 patients.

The randomization of the participants to be included in each group will be done using the software "Research Randomizer" (www.randomizer.org).

The randomization procedure will be performed by an independent research unrelated to the study. The randomization file will be saved in a password-protected online database. This independent research will enrol participants and will assign the patients to intervention groups.

Definition of study conclusion For each patient, the study is considered closed upon the discharge of from the rehabilitation unit.

Data analysis

Student's t-test and chi-square analyses were used to assess the differences between the demographic and clinical background characteristics of participants in the two conditions. The effects of the two treatments over time were assessed by repeated-measures analysis of variance, with one between-subjects factor (treatment) and one within subjects factor (time).

The investigators will measure the effects of the intervention on the power spectra of frequency band extracted from the EEG recordings, using MATLAB (Brainstorm, for the PSD analysis and EEGLab for the preprocessing of the EEG recordings) Data monitoring and management A data monitoring committee has not been necessary because the study is considered to be of minimal risk. The paper and pencil tests and questionnaire will be stored in a locked cabinet and will be entered in an electronic file. The access to these data will be permitted to the research members only.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Traumatic brain injury (TBI)
* Rancho Level of Cognitive Functioning (LCF) for TBI patients > 4
* Admission within 90 days from the onset

Exclusion Criteria:

* Unilateral Spatial Neglect
* Aphasia
* Severe vigilance deficits
* Severe verbal comprehension deficits
* Motor deficits of both hands
* Previous neurological stroke
* Previous neurological disease
* Previous psychiatric disease
* Use of alcohol or drugs
* Severe visual deficits
* Premorbid dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological primary outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Montreal Cognitive Assessment (MoCA) (0-30). High score means a better outcome.

SECONDARY OUTCOMES:
Neurophysiological secondary outcome | From the enrollment to the end of treatment at 2 weeks.
  The investigator will collect power spectra of frequency bands from continuous EEG resting state for 10 minutes (close+open eyes), before and after the treatment. EEGs were recorded with Ag/AgCl electrodes attached according to the 10-20 system.
  EEG data will be acquired, using a Galileo Mizar Plus medical device including 19 electrode channels (Fp1, Fp2,F7, F3, Fz, F4, F8, C3, Cz, C4, T7, T8, P7, P3, Pz, P4, P8, O1, O2), also during the last rehabilitation session. For obtaining the neurophysiological primary outcome measures, the invstigators will compute the power spectra of frequency bands from continuous EEG to assess the residual neuroplastic processes existing in patients, and the investigators will then evaluate the putative modulation of these processes by the combined intervention of prisms and serious games compared with traditional rehabilitation training.
Neuropsychiatric outcome | From the enrollment to the end of treatment at 2 weeks.
  - Neuropsychiatric Inventory (0-144): assesses 12 behavioral domains: delusions, hallucinations,agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, aberrant motor activity, night-time behavioral disturbances and appetite/eating disorders. The caregiver must rate the severity of the neuropsychiatric disturbances on a scale from 1 to 3, and the frequency from 1 to 4. High score means a worse outcome
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Stroop Test: this measures the ability to control and inhibit the automatic response. We used a short version of this test, with three tasks: (1) Word reading: the 30 stimuli are the written names of three colors (green, blue, and red). The subject must read the word as quickly as possible. (2) Color naming: 30 colored (green, blue, and red) circles are presented in a randomized order. The subject is asked to name the color of the circle. (3) Color naming of coloured words: 30 words (green, blue, and red) written in conflicting colors are presented. The subject has to name the character color of the word and not read the word itself aloud. High score both time and errors (0-30) means a worse outcome.
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  Trail Making Test (TMT): this test explores visual-conceptual and visual-motor tracking and is divided into two parts, A and B. In part A the subject must first draw lines to consecutively connect the numbers from 1 to 25; in part B the subject must alternately connect the numbers from 1 to 13 and the letters from A to N. Scoring is based only on time, i.e., the number of seconds used to complete the test. High score means a worse outcome
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Semantic Verbal Fluency (0-...): the patient was asked to say as many words as possible belonging to a given semantic category (colors, animals, fruits, and city) in 2 minutes. High score means a better outcome.
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Phonological Verbal Fluency (0-...): the patient is asked to produce as many words as possible beginningwith the letters F, A, and S in 1 minute. High score means a better outcome.
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Raven's Colored Progressive Matrices (0-36): the patient must logically complete a given visual spatial pattern, choosing from a set of six alternatives. This provides a nonverbal measure of intellectual ability. High score means a better outcome.
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Corsi span Backward (0-9): the same procedure is used for this test, but the subject has to reproduce the sequence of blocks in the reverse order. high score means a better outcome
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Digit span Backward (0-9): the same procedure is used for this test, but the subject has to reproduce the sequence of digit in the reverse order. High score means a better outcome
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Digit span Forward (0-9): the subject must repeat the lists of digits of increasing length immediately after presentation. The digit span score is the length of the longest correctly recalled sequence. High score means a better outcome
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Corsi span Forward (0-9): In a group of nine blocks the examiner taps some in a particular sequence then asks the patient to tap out exactly the same string immediately afterwards. Sequences of increasing length were presented. The spatial span score is the length of the longest sequence correctly recalled.
Neuropsychological outcome measure | From the enrollment to the end of treatment at 2 weeks.
  - Rey's 15-word Immediate (0-75) and Delayed Recall (0-15): the patient must recall a 15-word list, five times (immediate recall and learning); the sixth recall trial is performed 15 minutes later (delayed recall). High score means a better outcome.

OTHER OUTCOMES:
Functional cognitive secondary outcome | From the enrollment to the end of treatment at 2 weeks.
  For the assessment of functional outcome, the following scales will be used:
  - Functional Assessment Measure (FAM) cognitive subscale (14-98), composed of 14 items evaluating comprehension, expression, reading, writing, speech intelligibility, social interaction, emotional status, adjustment to limitation, employability, problem solving, memory, orientation, attention span and safety judgment. High score means a better outcome.
Functional secondary outcome | From the enrollment to the end of treatment at 2 weeks.
  The Modified version of Barthel Index (BI) (0-100): composed of 10 variables, describing activities of daily living and mobility. The maximum total score is 100 points depending on the autonomy of the patients in performing the sub-tasks of the scale. High score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simona Spaccavento, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS
Locations (4):
- Italy (4):
  - Istituti Clinici Scientifici Maugeri IRCCS, Bari
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia
  - Istituti Clinici Scientifici Maugeri IRCCS, Sciacca
  - Istituti Clinici Scientifici Maugeri IRCCS, Telese Terme

IPD SHARING:
Plan to Share IPD: Undecided